CLINICAL TRIAL: NCT03611647
Title: Correlating Probiotic Dietary Supplements During Pregnancy With Maternal Microbiome Profiles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Louise Laurent, MD/PhD, Director of Perinatal Research; Department of Obstetrics, Gynecology, and Reproductive Sciences; Division of Maternal-Fetal Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 171759
Record Dates: First submitted 2018-06-30; First posted 2018-08-02 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Pregnancy Related
Keywords: Microbiome; Probiotic
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Active Comparator)
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Probiotic dietary supplement containing a mixture of Lactobacillus and Bifidobacterium species, taken by mouth once daily for 4-6 weeks.
  Arms: Probiotic
Dietary Supplement: Placebo — Placebo, taken by mouth once daily for 4-6 weeks.
  Arms: Placebo

SUMMARY:
The overarching goal of this project is to compare the microbiome profiles of healthy pregnant women, both before and after the introduction of a probiotic supplement into the maternal diet. Specifically, the investigators are performing a pilot randomized double-blinded placebo-controlled trial, comparing the microbiome profiles of 40 healthy pregnant women randomized to receive an oral probiotic containing a mixture of Lactobacillus and Bifidobacterium species (20 mothers) versus an oral placebo (20 mothers) during the first/second trimester of pregnancy. For each mother, the investigators will collect biospecimens from the vagina, rectum, and urine, both before intervention, and 4-6 weeks after intervention. These biospecimens will be analyzed to obtain their microbiome profiles using next-generation sequencing. The primary outcome of interest is the vaginal microbiome, with secondary outcomes including the microbiomes of the rectum and urine. Additionally, the investigators will collect clinical data from the mother's and infant's medical records to correlate our findings with pregnancy and postnatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients ≥ 18 years of age
* Singleton pregnancy
* Gestational age 6 weeks and 0 days through gestational age 13 weeks and 6 days

Exclusion Criteria:

* Pregnant patients <18 years of age
* Multiple gestations
* Gestational age less than or equal to 5 weeks and 6 days
* Gestational age greater than or equal to 14 weeks and 0 days
* Institutionalization for psychiatric disorder, mental retardation, or criminal activity
* Inability to provide informed consent
* Major medical complication of pregnancy, including but not limited to: Diabetes, Chronic hypertension, Severe obesity with body mass index greater than or equal to 40 kg/m2
* Major surgical complications of pregnancy, including but not limited to: History of Bariatric surgery
* Major obstetrical complication of pregnancy, including but not limited to: History of spontaneous preterm birth
* Known maternal or fetal chromosomal abnormality
* Major fetal anomaly
* Intrauterine fetal demise
* Human immunodeficiency virus (HIV) or Hepatitis
* Chronic immunosuppressive medications or steroids
* Current use of probiotic supplementation
* Active urinary or vaginal infection
* Current use of antibiotics
* Current use of vaginal medication (e.g. vaginal progesterone)
* Cerclage in place

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Vaginal Microbiome, 16S rRNA | Baseline, and 4-6 weeks after intervention

SECONDARY OUTCOMES:
Change in Rectal Microbiome, 16S rRNA | Baseline, and 4-6 weeks after intervention
Change in Urinary Microbiome, 16S rRNA | Baseline, and 4-6 weeks after intervention

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - UCSD, La Jolla Clinic, 8910 Villa La Jolla Drive, La Jolla, California
  - UCSD, Hillcrest Clinic, Medical Offices South, San Diego, California
  - UCSD, Sorrento Valley Clinic, Directors Place, San Diego, California

IPD SHARING:
Plan to Share IPD: No